CLINICAL TRIAL: NCT06130137
Title: Genome-based Multiomics Analysis on Gut Microbiome in People Living With HIV and HBV
Brief Title: Gut Microbiome in People Living With HIV and HBV
Status: Not yet recruiting | Type: Observational
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Kyunghee University Medical Center (Other); Hanyang University (Other)
Responsible Party: Principal Investigator, Eun-Jeong Joo, M.D, Ph.D, Kangbuk Samsung Hospital
Other Study IDs: HIVHBVgutmicrobiome
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Human Immunodeficiency Virus; Chronic Hepatitis b; Gut Microbiome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV: Patients with HIV infection
- HBV: Patients with HBV infection

SUMMARY:
Building a Microbiome Data Platform and Conducting Clinical Evidence Research in Individuals Infected with the Human Immunodeficiency Virus (HIV) and Hepatitis B virus.

DETAILED DESCRIPTION:
Chronic HIV infection, which often results in metabolic disorders, leads to shifts in the gut microbiota, contributing to immune activation and chronic inflammation. This study seeks to compare the gut microbiota in individuals with chronic HIV infection and chronic hepatitis B patients. The objective is to identify specific gut bacterial strains and metabolic pathways linked to the metabolic disorders commonly observed in HIV patients.

ELIGIBILITY:
Inclusion Criteria:

1. HIV patients

   * Inidividuals over 19 years old
   * HIV patients on antiretroviral therapy (ART)
2. HBV patients

   * Individuals over 19 years old
   * Chronic hepatitis B patients with either chronic hepatitis, liver cirrhosis or hepatocellular carcinoma

Exclusion Criteria:

1. Patients with indeterminate colitis
2. Individuals who have used antibiotics or steroids within 24 hours of the microbiome sample collection (excluding antiviral treatments for hepatitis B and HIV)
3. Individuals who have used vaginal or external medications, including antifungal agents, within 24 hours of microbiome sample collection
4. Those with acute illnesses, with or without fever, of moderate or severe severity; however, sampling may be postponed until the subject recovers.
5. Individuals with gastrointestinal disorders that may impact microbiome analysis and are currently medically uncontrolled or under treatment for the respective condition
6. Individuals with a positive result in a urine pregnancy test, pregnant, or breastfeeding at the time of microbiome sample collection
7. Individuals for whom medical opinions suspect that they may have an impact on the sample collection at the time of microbiome collection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic viral diseases will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect clinical information data and stool from HIV and HBV patients | 2 years
  Clinical information data will be collected from both HIV and HBV infected patients. Biosamples collected from these individuals will be used to establish a multi-omics analysis platform, including the examination of the intestinal microbiome. With this platform, comparative clinical studies will be conducted to uncover the disease's pathophysiology and identify potential biomarkers related to metabolic diseases.

SECONDARY OUTCOMES:
Shotgun metagenomic sequencing will be done with stool collected from HIV and HBV patients | 2 years
  Diversity analysis: Alpha and beta diversity analyses are conducted to determine differences in the composition of gut microbiota between healthy individuals and patients.
  Important feature selection: Differential abundance analysis (e.g., using methods like LEfSe or ANCOM) or machine learning (e.g., random forest, support vector machine) is employed to identify microbiota.
  Functional profile prediction: In cases where metagenomic analysis is not feasible, the PICRUSt2 program is utilized to predict and analyze functional profiles based on the phylogeny of the microbiota present in healthy individuals and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eunjeong Joo, M.D., Ph.D, Principal Investigator — Kangbuk Samsung Hospital

IPD SHARING:
Plan to Share IPD: No